CLINICAL TRIAL: NCT01406886
Title: Combined Effects of Energy Density and Eating Rate on Energy Intake and Biomarkers of Satiety
Brief Title: Combined Effects of Energy Density and Eating Rate on Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Principal Investigator, James Philip Karl, Research Dietitian, United States Army Research Institute of Environmental Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: H09-28
Record Dates: First submitted 2011-07-05; First posted 2011-08-01 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Appetite
Keywords: Modifiable environmental; behavioral factors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Energy density (Experimental): Low or high energy density meal
  Interventions: Behavioral: Eating rate

INTERVENTIONS:
Behavioral: Eating rate

SUMMARY:
This study will examine the independent and combined effects of energy density and eating rate on appetite and endocrine mediators of appetite. Increasing eating rate and energy intake are expected to additively increase energy intake.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-27 kg/m2
* Weight stable

Exclusion criteria:

* Chronic used of OTC or prescription drugs known to affect metabolism
* Chronic disease
* Gastric bypass surgery
* Disordered eating
* Pregnant or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Energy intake | 1 meal

SECONDARY OUTCOMES:
Subjective appetite | 0-180 min
Postprandial peptide-YY response | 0-180 min
Postprandial ghrelin response | 0-180 min
Postprandial glucagon-like peptide-1 response | 0-180 min
Postprandial pancreatic polypeptide response | 0-180 min

CONTACTS AND LOCATIONS:
Overall Officials: Scott J Montain, PhD, Principal Investigator — US Army Research Institute of Environmental Medicine
Locations (1):
- USARIEM, Natick, Massachusetts, United States

REFERENCES:
- [Result] Karl JP, Young AJ, Rood JC, Montain SJ. Independent and combined effects of eating rate and energy density on energy intake, appetite, and gut hormones. Obesity (Silver Spring). 2013 Mar;21(3):E244-52. doi: 10.1002/oby.20075. PMID 23592679